CLINICAL TRIAL: NCT00469911
Title: Quantification of Intramyocardial Lipid by Proton Magnetic Resonance Spectroscopy
Acronym: MRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5P20RR02064302; 05-0759 (Other: HRPO); P20RR020643 (NIH)
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Heart Transplantation
Keywords: Heart; Transplant; MRS; MRI; Spectroscopy
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Compare magnetic resonance imaging measurements of triglyceride accumulation in myocardial tissue with ex vivo myocardial tissue collected from heart transplant patients who have had routine clinical heart biopsy.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnetic Resonance Spectroscopy (Experimental): Patients will have Magnetic Resonance Spectroscopy to measure in vivo accumulation of triglycerides in myocardial tissue
  Interventions: Procedure: Magnetic Resonance Spectroscopy
- Ex vivo heart biopsy (Experimental): Patients will have their normal routine clinical heart biopsy of myocardial heart tissue.
  Interventions: Procedure: Ex vivo heart biopsy

INTERVENTIONS:
Procedure: Magnetic Resonance Spectroscopy — Magnetic Resonance Spectroscopy is a noninvasive procedure that provides detailed body images on any plane.
  Other Names: MRS
  Arms: Magnetic Resonance Spectroscopy
Procedure: Ex vivo heart biopsy — Heart transplant patients will have their normal clinical routine heart biopsy
  Other Names: heart biopsy
  Arms: Ex vivo heart biopsy

SUMMARY:
Accumulation of triglycerides in heart tissue has been associated with changes in left ventricular function which can lead to heart failure. Proton magnetic resonance spectroscopy is currently the only non-invasive in vivo method to measure myocardial triglycerides content. The primary goal of this study was to determine if Magnetic Resonance Spectroscopy could effectively measure myocardial triglyceride content in myocardial heart tissue. Thus, quantitative and reliable techniques to monitor in vivo triglyceride accumulation in the heart are important for disease diagnosis and management. Currently, no such imaging method exists.

DETAILED DESCRIPTION:
Because routine biopsy of the myocardium is not feasible, MRS is the most promising technique for the quantification of myocardial triglycerides. MRS is routinely used to precisely characterize metabolite concentrations in muscle and liver. 14-16 Studies such as monitoring the levels of deoxymyoglobin and real-time tracking of the postprandial accumulation of cellular lipids are examples of its diversity and potential.15,17,18 Generally, these studies suggest that the reproducibility of MRS is between 2 and 6%.18,19 In vivo cardiac MRS provides unique challenges because of the requirement to compensate for concurrent heart and lung motion. Using cardiac and respiratory gating to minimize motional artifacts, an initial validation study found a variation of 17% for sequential measurements, attributing the major error to residual motional effects. 20 Moreover, measurements were limited to the inter-ventricular septum. Using navigator and cardiac gating appeared to give a slight, 4%, improvement, but this was a preliminary study and no validation was done.21 For a comprehensive clinical validation, other reproducibility factors must be addressed. Variations due to post-processing, coil placement and calibration, trigger reproducibility, internal versus external standard, shimming, and protocol sequence variables such as pulse quality, gradient strength, voxel size, relaxation time, echo time, and the number of scan repetitions are all known sources of reproducibility. 17,19,22-24 All of these variables must be characterized in order to achieve optimal inter- scanner and subject reproducibility along with accurate treatment tracking capability. Therefore, 10 normal healthy volunteers were imaged to determine the reliability of the MRS protocol with test-re-test measurements. The 8 heart transplant patients were imaged prior to their routine heart biopsies, and then the myocardial biopsy tissue was measure and compared to the pre-biopsy images.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* heart transplant patients
* undergoing post transplant endomyocardial biopsy
* not experiencing significant rejection
* heart transplant patients must be 18-30 years old.

Exclusion Criteria:

* <18 or >45
* pregnant
* significant systemic illness
* actively ill
* acute transplant rejection
* any condition that would prevent a participant from completing the NMR spectroscopy (i.e pacemakers, claustrophobia)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gropler, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Medical School, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kannel WB, McGee DL. Diabetes and cardiovascular disease. The Framingham study. JAMA. 1979 May 11;241(19):2035-8. doi: 10.1001/jama.241.19.2035. PMID 430798
- [Background] Koskinen P, Manttari M, Manninen V, Huttunen JK, Heinonen OP, Frick MH. Coronary heart disease incidence in NIDDM patients in the Helsinki Heart Study. Diabetes Care. 1992 Jul;15(7):820-5. doi: 10.2337/diacare.15.7.820. PMID 1516498
- [Background] Abbott RD, Donahue RP, Kannel WB, Wilson PW. The impact of diabetes on survival following myocardial infarction in men vs women. The Framingham Study. JAMA. 1988 Dec 16;260(23):3456-60. PMID 2974889
- [Background] Kannel WB, Hjortland M, Castelli WP. Role of diabetes in congestive heart failure: the Framingham study. Am J Cardiol. 1974 Jul;34(1):29-34. doi: 10.1016/0002-9149(74)90089-7. No abstract available. PMID 4835750
- [Background] Zhou YT, Grayburn P, Karim A, Shimabukuro M, Higa M, Baetens D, Orci L, Unger RH. Lipotoxic heart disease in obese rats: implications for human obesity. Proc Natl Acad Sci U S A. 2000 Feb 15;97(4):1784-9. doi: 10.1073/pnas.97.4.1784. PMID 10677535

RESULTS

PARTICIPANT FLOW:
Groups:
- Heart Transplant: Compare Magnetic resonance myocardial lipid measurements with biopsy derived ex vivo measurements
  Magnetic Resonance Spectroscopy: It is basically the same as an MRI. It is a noninvasive procedure that provides detailed body images on any plane.
  Endocardial Biopsy: This is a standard of care procedure that is already performed on heart transplant patients. This is a procedure that takes a biopsy (tissue sample) of the heart muscle.
- Controls: Normal volunteers used to assess reproducability of the MRS measurements
Period: Overall Study
Arm/Group | Heart Transplant | Controls
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Heart Transplant: Compare Magnetic resonance myocardial lipid measurements with biopsy derived ex vivo measurements
  Magnetic Resonance Spectroscopy: It is a noninvasive procedure that provides detailed body images on any plane.
  Endocardial Biopsy: This is a standard of care procedure that is already performed on heart transplant patients. This is a procedure that takes a biopsy (tissue sample) of the heart muscle.
- Control Subjects: Control subjects with a broad range of body mass indexes and physiological conditions.
- Total: Total of all reporting groups
Arm/Group | Heart Transplant | Control Subjects | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 10 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Correlation Co-efficient Between MRS Spectroscopy and Endomyocardial Biopsy in Heart Transplant Participants
Description: Participants first had MRS spectroscopy then the MRS spectroscopy images were compared to endomyocardial biopsy
Time Frame: 2 to 10 days
Measure: Number; unit: correlation co-efficient
Groups:
- Heart Transplant Patients: Measurement of triglycerides in heart transplant patients using MRI
Arm/Group | Heart Transplant Patients
Number analyzed (Participants) | 8
correlation co-efficient | 0.97
Statistical Analysis 1: Comparison: Heart Transplant Patients; Test type: Superiority; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 to 10 days
Groups:
- Heart Transplant - Endomyocardial Biopsy: This is a procedure that takes a biopsy (tissue sample) of the heart muscle., and it was compared to the MRS Spectroscopy images
- Control Subjects: Normal volunteers used to assess reproducability of the MRS measurements
Arm/Group | Heart Transplant - Endomyocardial Biopsy | Control Subjects
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

LIMITATIONS AND CAVEATS:
There were no limitations or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes